CLINICAL TRIAL: NCT01939470
Title: Oklahoma Native American Women's Osteoporosis Screening Study
Status: Completed | Type: Observational
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Other Study IDs: HE0840
Record Dates: First submitted 2013-08-01; First posted 2013-09-11 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis
Keywords: osteoporosis; bone; inflammation; diabetes; vitamin D
MeSH Terms: conditions — Osteoporosis; Inflammation; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Native American Women: Native American Women over the age of 50 yrs

SUMMARY:
Native American women may be considered high risk for osteoporosis due to lifestyle factors and incidence of type 2 diabetes. The objectives of this study are to: 1) determine the prevalence of osteopenia/osteoporosis in Native American female volunteers; 2) to evaluate their rate of bone loss; 3) to assess the relationship between lifestyle factors, inflammatory mediators, and select endocrine parameters on osteoporosis risk; and 4) determine the barriers to treatment. Participants will undergo a baseline, Year 1 and Year 2 follow-up osteoporosis risk assessment. Data will be analyzed using repeated measures ANOVA and logistical regression.

DETAILED DESCRIPTION:
Osteoporosis, characterized by decreased bone density and deterioration in bone microarchitecture, is estimated to afflict 1 out of 2 women over the age of 50 years. These estimates are based primarily on Caucasian populations with limited information in Native Americans. Native American women may be considered high risk for osteoporosis due to lifestyle factors in conjunction with the incidence of diabetes. The objectives of this study are to: 1) determine the prevalence of osteopenia/osteoporosis in Native American female volunteers, aged 50+ years, who are eligible for health care through Indian Health Services; 2) to evaluate their rate of bone loss, 3) to assess the relationship between lifestyle factors, inflammatory mediators, and select endocrine parameters on osteoporosis risk; and 4) determine the barriers to treatment. Native American women aged, 50+ years, who are eligible for services through Indian Health Services in the Oklahoma City (OKC) Area will be recruited. Participants will undergo a baseline osteoporosis risk assessment, i.e. medical history, dual-energy x-ray absorptiometry (DXA) scans, dietary and physical activity assessment, and optional blood draw, and then encouraged to return to their primary care physician for counsel and/or treatment. Serum markers of bone metabolism, endocrine parameters (e.g. vitamin D metabolites) and inflammatory molecules will be assessed for participants that consent to the blood draw. All participants will receive educational information related to osteoporosis risk and prevention, and follow-up visits scheduled at the end of Year 1 and Year 2. Data will be analyzed using repeated measures ANOVA and logistical regression with the α set at 0.05 for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Native American women who are eligible fore services at Indian Health Clinics in OKC
* 50 years of age or older

Exclusion Criteria:

* Women who weigh more than 300 lbs or who are pregnant or cognitively impaired

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample of Native American who are eligible for health care services at Indian Health Clinics in the Oklahoma City area
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Bone Mineral Density at Year 1 and Year 2 | Baseline, year 1 and year 2

SECONDARY OUTCOMES:
Change from Baseline in Serum Bone Formation Markers (bone-specific alkaline phosphatase) at Year 1 and Year 2 | Baseline, year 1 and year 2
Change from Baseline in Bone Resorption Markers (C-telopeptide) at Year 1 and Year 2 | Baseline, year 1 and year 2
Change from Baseline in Serum 25-Hydroxy Vitamin D at Year 1 and Year 2 | Baseline, year 1 and year 2
Change from Baseline in Serum Interleukin-6 at Year 1 and Year 2 | Baseline, year 1 and year 2
Change from Baseline in C-reactive Protein at Year 1 and Year 2 | Baseline, year 1 and year 2

CONTACTS AND LOCATIONS:
Overall Officials: Brenda J. Smith, Ph.D., Principal Investigator — Oklahoma State University
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States